CLINICAL TRIAL: NCT03521479
Title: A Phase 2, Muti-Center Study of Repeat Dosing of Squaric Acid Dibutyl Ester in Subjects With Herpes Labialis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug out of specification
Sponsor: Squarex, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P2c
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Herpes Labialis; HSV
Keywords: Squaric Acid; SADBE; Squaric acid dibutyl ester
MeSH Terms: conditions — Herpes Labialis | interventions — squaric acid dibutyl ester

STUDY DESIGN:
Intervention Model Description: Subjects will receive on a double blind basis one of two treatment regimens:
  * Group A: 15 subjects, treated with 2% SADBE on day 0 and with 2% SADBE on the visits at week 3, week 6, week 9, and month 8.
  * Group B: 15 subjects, treated with 2% SADBE on day 0 and with 0.5% SADBE on the visits at week 3, week 6, week 9, and month 8.
  And subjects will be recruited on an open label basis to two other treatment regimens:
  * Group C: 15 subjects, treated with 2% SADBE on day 0, month 3, and month 6.
  * Group D: 15 subjects, treated with 2% SADBE on day 0 and month 6.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The double-blinding only applies between groups A and B. Subjects for groups C and D will be recruited on an open label basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Treated with 2% Squaric Acid Dibutyl Ester (SADBE) on day 0 and with 2% SADBE on the visits at week 3, week 6, week 9, and month 8.
  Interventions: Drug: Squaric Acid Dibutyl Ester
- Group B (Experimental): Treated with 2% Squaric Acid Dibutyl Ester (SADBE) on day 0 and with 0.5% SADBE on the visits at week 3, week 6, week 9, and month 8.
  Interventions: Drug: Squaric Acid Dibutyl Ester
- Group C (Active Comparator): Treated with 2% Squaric Acid Dibutyl Ester (SADBE) on day 0, month 3, and month 6.
  Interventions: Drug: Squaric Acid Dibutyl Ester
- Group D (Active Comparator): Treated with 2% Squaric Acid Dibutyl Ester (SADBE) on day 0 and month 6.
  Interventions: Drug: Squaric Acid Dibutyl Ester

INTERVENTIONS:
Drug: Squaric Acid Dibutyl Ester — Repeat topical application of 2% and 0.5% squaric acid dibutyl ester (SADBE) in subjects with frequent herpes labialis (4 or more episodes in the previous 12 months).
  Other Names: Repeat Dosing

SUMMARY:
Primary Objective: To assess local and generalized adverse events with repeat topical application of 2% and 0.5% squaric acid dibutyl ester (SADBE) in subjects with frequent herpes labialis (4 or more episodes in the previous 12 months).

Secondary Objective: To assess efficacy of repeat topical application of 2% and 0.5% SADBE in the prevention of herpes labialis episodes.

DETAILED DESCRIPTION:
Primary oral infection with the herpes simplex virus (HSV) typically occurs at a young age, is asymptomatic, and is not associated with significant morbidity. After primary oral infection, HSV may persist in a latent state in the trigeminal ganglion and later reactivate as the more common herpes labialis, or "cold sores." Common triggers for reactivation are well known and include ultraviolet light, trauma, fatigue, stress, fever, inflammation, and menstruation. These lesions affect up to 45 percent of the U.S. population. They classically manifest as a well-localized cluster of small vesicles along the vermilion border of the lip or adjacent skin. The vesicles subsequently rupture, ulcerate, and crust within 24 to 48 hours. Spontaneous healing occurs over seven to 10 days.

In immunocompetent patients, herpes labialis usually is mild and self-limited. However, pain, swelling, and cosmetic concerns may prompt physician consultation. Orally administered antiviral agents, such as acyclovir (Zovirax) or valacyclovir (Valtrex), have a modest clinical benefit if initiated during the prodrome. Topical treatment with 1% penciclovir cream (Denavir) may reduce healing time and pain slightly, even if initiated after the prodrome. However, reduction in healing time with systemic or topical agents is modest.

Squaric acid dibutyl ester (SADBE) is a topical immunotherapeutic agent used in the treatment of verruca vulgaris and alopecia areata. During a recent FDA Compounding Advisory Committee Meeting, it was recommended that squaric acid dibutylester be included on the list of bulk drug substances allowed for use in compounding under section 503A of the Federal Food, Drug, and Cosmetic Act. And SADBE has now been so listed under section 503A.

A study completed by Lee et al of 29 patients with recalcitrant warts demonstrated complete clearance in 69% of patients with application every 2-4 weeks. Silverberg et al showed a complete clearance in 58% of patients (n=61) when SADBE was applied 3 times weekly. A placebo-controlled clinical study completed at Massachusetts General Hospital showed that squaric acid prevented recurrence of herpetic lesions. The effect of SADBE of delaying new herpes labialis outbreaks was highly significant (p<0.01) as compared to placebo.

Primary Objective: To assess local and generalized adverse events with repeat topical application of 2% and 0.5% squaric acid dibutyl ester (SADBE) in subjects with frequent herpes labialis (4 or more episodes in the previous 12 months).

Secondary Objective: To assess efficacy of repeat topical application of 2% and 0.5% SADBE in the prevention of herpes labialis episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 65
2. Clinical diagnosis of herpes labialis, which may be made at the screening visit based on the patient's self-reported history of symptoms. An active herpes labialis outbreak at the time of entry into the clinical trial will neither be required nor will be an exclusion criterion.
3. Self report having four (4) or more episodes of herpes labialis in the past 12 months.

   Subjects will NOT be told that four-or-more episodes in the previous 12 months is the entry criterion. Subjects will be asked "How many separate episodes of cold sores have you had in the previous 12 months?" They will be included if they give an answer of four or more and excluded if they give an answer of three or fewer.
4. At least half of the subject's episodes of the previous 12 months should be vesicular in nature and at least half preceded by prodromal symptoms. Prodromal symptoms may include tingling, itching, burning or pain before the development of a herpetic lesion.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Current or recurrent non-herpetic infection or any underlying condition that may predispose to infection or anyone who has been admitted to the hospital due to bacteremia, pneumonia or any other serious infection in the last 12 months.
3. Therapy with glucocorticoid or immunosuppressants at time of recruitment or within past 4 weeks prior to the screening visit, or at any time during the study (including inhaled corticosteroids for asthma), except for topical steroids in sites other than face.
4. History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers).
5. History of organ transplantation.
6. HIV-positive status determined by history at screening or known history of any other immunosuppressive disease.
7. Severe co-morbidities (CHF [NYHA class II or worse], MI, CVA or TIA) within 3 months of screening visit, current unstable angina pectoris or oxygen-dependent severe pulmonary disease.
8. Known hypersensitivity to Dimethyl sulfoxide (DMSO).
9. Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.
10. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of the screening visit.
11. Previous exposure to SADBE (squaric acid or squaric acid dibutyl ester).
12. Subject has an abnormal skin condition (e.g., acne, eczema, rosacea, psoriasis, albinism, or chronic vesiculo-bullous disorder) that occurs in the area ordinarily affected by herpes labialis
13. Subject has an abnormal skin condition (e.g., eczema, rosacea, psoriasis, albinism, or chronic vesiculo-bullous disorder) that occurs in the inner aspect of either upper arm (the area where drug will be applied).
14. Subject has had a vaccine for either HSV-1 or HSV-2.
15. Subject has had treatment with anti-viral therapy (including ABREVA) within 2 weeks before first dose of SADBE or at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - International Research Partners, LLC, Doral, Florida
  - Prism Clinical Research, LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.3) | 39.2 (10.1) | 47.1 (12.4) | 47.2 (13.1) | 43.94 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 6 | 23
  Male | 3 | 5 | 5 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 2
  African American or Black | 0 | 0 | 1 | 1 | 2
  White | 8 | 9 | 7 | 8 | 32
  Hispanic or Latino | 1 | 0 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Local and Generalized Adverse Events
Description: Local and generalized adverse events with repeat topical application of 2% and 0.5% squaric acid dibutyl ester (SADBE) in subjects with frequent herpes labialis (4 or more episodes in the previous 12 months).
Time Frame: 9 months
Measure: Number; unit: events
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 10 | 10 | 10 | 10
events
  Localized reaction (rash, erythema, itching/pruritus, warmth/burning) at application site | 24 | 14 | 17 | 6
  Generalized adverse events (related, possible or greater) | 2 | 3 | 1 | 0
  Generalized adverse event (unrelated) | 4 | 7 | 6 | 4

ADVERSE EVENTS:
Time Frame: 172 days
Description: At risk participants listed below as 30 because the 10 participants in each group was counted on 3 separate occasions.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 13/30 | 12/30 | 6/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group A (N=30) | Group B (N=30) | Group C (N=30) | Group D (N=30)
Rash (Skin and subcutaneous tissue disorders) | 3/10 | 6/10 | 6/10 | 4/10 — Day 0-20
Rash (Skin and subcutaneous tissue disorders) | 6/10 | 6/10 | 0/10 | 0/10 — Day 21-41
Rash (Skin and subcutaneous tissue disorders) | 4/10 | 0/10 | 0/10 | 0/10 — Day 42+

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03521479/Prot_SAP_000.pdf